CLINICAL TRIAL: NCT02412397
Title: DePuy Global Unite Shoulder System
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Rothman Institute Orthopaedics (Other)
Responsible Party: Sponsor
Other Study IDs: 15Jabb
Record Dates: First submitted 2015-04-06; First posted 2015-04-09 (Estimated); Last update posted 2015-04-09 (Estimated); Status verified 2015-04

CONDITIONS: Osteoarthritis
Keywords: Shoulder
MeSH Terms: conditions — Osteoarthritis | interventions — Arthroplasty, Replacement, Shoulder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional

INTERVENTIONS:
Procedure: Total Shoulder Arthroplasty

SUMMARY:
To collect medium to long-term survivorship implant outcomes on the DePuy Global Unite Shoulder System

ELIGIBILITY:
Inclusion Criteria:

* Patient greater than 18 years of age and skeletally mature
* Patient qualifies for primary or revision total or reverse shoulder arthroplasty based on diagnosis of investigator of osteoarthritis, rheumatoid arthritis, post-traumatic arthritis, un-united humeral head fractures, irreducible 3- and 4- part proximal humeral fracture, avascular necrosis, or gross rotator cuff deficiency.
* Patient is willing and able to provide written informed consent and to complete scheduled follow up visits/evaluations/questionnaires

Exclusion Criteria:

* Patient has one of the following compromise the affected limb; a significant injury to the upper brachial plexus, paralysis of the axillary nerve, or a neuromuscular disease compromising the affected limb
* Patient has a known or suspected infection
* Patient is known to be pregnant
* Patient has a sensitivity or allergic reaction to one or more of the implanted materials
* Patient is unwilling or unable to provide consent or comply with follow up visits

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients who were implanted with the DePuy Global Unite Shoulder System
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Primary Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Implant Survivorship | 10 years post-operative